CLINICAL TRIAL: NCT03902977
Title: Effect of Quilting Sutures on Post-operative Drainage After Mastectomy and/or Axillary Lymph Node Dissection in Patients With Breast Cancer: a Single Blind Randomised Phase III Controlled Trial
Brief Title: Effect of Quilting Sutures on Post-operative Drainage After Mastectomy and/or Axillary Lymph Node Dissection
Acronym: Quilting
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient recruitment
Sponsor: Lindenhofgruppe AG (Industry)
Collaborators: University of Bern (Other); StiftungLindenhof (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BZ01/17; 17-17-F (Other: StiftungLindenhof)
Record Dates: First submitted 2019-03-25; First posted 2019-04-04 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Intervention Model Description: All patients have undergone surgery for treatment of breast cancer. During surgery they are assigned to one of two groups (randomization 1:1): quilting or conventional suture.
Who Masked: Participant, Care Provider
Masking Description: The surgeon who operates the patient will neither perform the follow up visits nor contact other investigators. A blinded investigator will see the patient at the following visits after surgery: week 1, week 4 and week 12. In case the patient develops a seroma which needs aspiration, aspiration will be performed by the blinded investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): quilting
  Interventions: Procedure: quilting
- Arm B (Active Comparator): conventional suture
  Interventions: Procedure: conventional suture

INTERVENTIONS:
Procedure: quilting — After mastectomies or ALND dissections using standard technique for wound closure multiple sutures (monocryl 3.0) every 3 to 4 cm in the site of the mastectomy (1 or 2 rows) or in the dissected axilla.Placement of one drain into the breast and axilla or in the axillary cavity by a separate stab incision
  Arms: Arm A
Procedure: conventional suture — After mastectomies or ALND dissections standard technique for wound closure. Placement of one drain into the breast and axilla or in the axillary cavity by a separate stab incision
  Arms: Arm B

SUMMARY:
Breast cancer is the most frequent type of cancer among Swiss women (5'700 cases diagnosed every year). Mastectomy is indicated when breast conservative surgery is not possible or by patient wish. Axillary lymph nodes dissection (ALND) is indicated primarily for node-positive breast cancer.

Postoperative seroma after mastectomy and axillary clearance is a common complication, occurring in 25 to more than 60% of patients with breast cancer. After mastectomy and/or ALND conventional wound closure commonly uses suction drain to prevent seroma. However, seroma frequently occurs after drain removal. Excessive fluid accumulation in seroma stretches the skin, resulting in patient discomfort, impaired ipsilateral shoulder function and higher risk of surgical site infection and prolongs the hospitalization. In rare cases, a fibrous encapsulated seroma is resistant to conservative treatment and requires surgical resection. Thus, seroma may also impact health care costs requiring longer hospital stay or unplanned outpatient visits and may delay adjuvant therapy.

Recent data suggest that quilting suture through flap fixation reduces the incidence of seroma. Therefore, quilting suture has the potential to increase patients' quality of life, as well as to shorten the length of hospital stay and to reduce hospital costs, providing the rationale for this study.The aim of our project is to compare the efficacy of quilting suture with that of conventional closure without quilting in reducing the drainage quantity, the length of hospitalisation and the prevalence of seroma following mastectomy and/or axilla for breast cancer, as well as the patient reported pain increasing patient quality of life.

The final goal is the omission of axillary drainage in the future. All randomised patients will be followed for 12 weeks. Patients will fill in 2 questionnaires (EQ5-D: European Quality of Life and Brief Pain Inventory: BPI). The Health Economic Analysis form (HEA) will be completed by the investigator collecting the patient data.

Total duration of study: 2.5 years. There are 2 treatments groups 50% of the study participants will be treated with quilting suture and 50% with conventional closure. Patients are randomly divided into the 2 groups. All patients are blinded to the surgical treatment.This means that they do not know which surgical treatment they have received (quilting suture or conventional closure), The operating surgeon will not see the after the operation. Seroma assessment will be performed by other medical personnel, that do not know which surgical treatment has been given. In case of seroma a physician (not the operating surgeon) will perform the aspiration of seroma if needed.

DETAILED DESCRIPTION:
Breast cancer is the most frequent type of cancer among Swiss women (5'700 cases diagnosed every year). Mastectomy is indicated when breast conservative surgery is not possible or by patient wish. Axillary lymph nodes dissection (ALND) is indicated primarily for node-positive breast cancer.

Postoperative seroma after mastectomy and axillary clearance is a common complication, occurring in 25 to more than 60% of patients with breast cancer. After mastectomy and/or ALND conventional wound closure commonly uses suction drain to prevent seroma. However, seroma frequently occurs after drain removal. Excessive fluid accumulation in seroma stretches the skin, resulting in patient discomfort, impaired ipsilateral shoulder function and higher risk of surgical site infection and prolongs the hospitalisation. In rare cases, a fibrous encapsulated seroma is resistant to conservative treatment and requires surgical resection. Thus, seroma may also impact health care costs requiring longer hospital stay or unplanned outpatient visits and may delay adjuvant therapy.

Recent data suggest that quilting suture through flap fixation reduces the incidence of seroma. Therefore, quilting suture has the potential to increase patients' quality of life, as well as to shorten the length of hospital stay and to reduce hospital costs The aim of this trial is to compare the efficacy of quilting suture of the dead space at the pectoral area and/or axilla with that of conventional suture in reducing the total volume of post-mastectomy and/or axillary drainage and seroma in female patients after surgical treatment of breast cancer.The study seeks primarily to determine if quilting suture compared to conventional suture after mastectomy/ALND reduces the total volume of axillary drainage until drain removal.

This single blind randomised phase III controlled superiority trial compares 2 surgical techniques: quilting suture and conventional suture. Patients will be assigned to one of 2 parallel groups: Arm A: quilting suture and Arm B: (no quilting suture): conventional wound closure.

Duration of accrual: 2 years - Duration of trial treatment: 1 day (surgery). Surgery procedure: Mastectomies or ALND dissections using a standardized technique, with multiple quilting sutures in the site of the mastectomy/in the dissected axilla or conventional closure without quilting. In both procedures placement of one drain into the breast and axilla or in the axillary cavity.

All randomised patients will be followed for 12 weeks. Patients will fill in 2 questionnaires (Quality of Life: EQ5-D and Brief Pain Inventory: BPI). The Health Economic Analysis form (HEA) will be completed by the investigator collecting the patient data.

At the study visits the following examinations will be performed: physical examination, blinded assessment of seroma, axillary drain volume, adverse events and surgical site infections.

The sample size is based on the primary endpoint, the total volume of axillary drainage. We assume a reduction in the total volume of axillary drainage of 200 ml in the intervention arm (application of quilting sutures) compared to the control arm (no application of sutures), which is based on literature and actual measurements in 14 patients. A total of 106 patients (53 in each group) will yield a power of 80% to detect this difference at a two-sided significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years-old female patients
* mastectomy alone, mastectomy and sentinel, mastectomy and axilla, axilla and tumorectomy or axilla alone
* patients with histo- or cytology proven breast cancer Union for International Cancer Control's (UICC)/American Joint Committee on Cancer (AJCC) stage I-III
* Fluency in either German or French
* The EQ-5D and BPI questionnaires must be completed by the patient at registration
* Patient has given written informed consent before registration.

Exclusion Criteria:

* Bilateral operation or reconstruction
* Psychiatric disorder precluding understanding of information on trial related topics, giving informed consent and/or filling out the questionnaires
* Pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Total volume (ml) of axillary/breast drainage until drain removal. | up to 5 days
  Blinded daily measurement of axillary drainage volume during hospital stay at 8.00 h a.m in the morning through nurses.

SECONDARY OUTCOMES:
Total duration (days) of breast/axillary drainage | 1-5 days
  calculated from the date of surgery to date of drain removal calculated drainage from the date of surgery to the date of axillary/breast drain removal
Duration of postoperative hospital stay | 5-7 days
  calculated from the date of surgery to the date of discharge (after surgery patients are hospitalized usually for 5 days)
Number of patients with clinically relevant seroma | From the date of surgery until 12 weeks after surgery
  Clinically relevant seroma is defined as either causing strong discomfort or requiring aspiration
Number of patients with lymphedema | From the date of surgery until week 12
  increase of more than 2.5 cm in arm circumference
Adverse Events (AEs) due to surgical procedure | during 4 weeks after surgery
  after surgery possible wound-related complications (e.g. haematoma requiring reoperation, skin flap necrosis) flap necrosis)
Surgical morbidity | within the 12 weeks follow up after surgery
  number of outpatient visits (related to mastectomy/ALND) needed following participant's discharge
Duration (number of days) of clinically relevant seroma aspiration period | from the date of surgery until 12 weeks after surgery
  calculated until the date of the last clinically relevant seroma aspiration
Volume of axillary drainage per 24 hours in ml | up to 5 days
  calculated as the total volume of axillary drainage in ml until drain removal divided by the total duration of axillary drainage in days
Number of clinically relevant seroma aspirations | From the date of surgery until 12 weeks after surgery
  Aspiration is performed if the patient experiences strong discomfort, in case of impaired ipsilateral shoulder function, if higher risk of surgical infection and in case pain interferences with daily functions
Total volume in ml of all clinically relevant seroma aspirations | From the date of surgery until 12 weeks after surgery
  calculated in in ml
Surgical morbidity | up to 2 hours
  intraoperative blood loss calculated in ml from start to end of surgery
Surgical morbidity | up to 2 hours
  duration of the surgical procedure from start to end of surgery

OTHER OUTCOMES:
Patient self-reported pain will be assessed with the Brief Pain Inventory (BPI) patient self-reported questionnaire | every day during the first 2 weeks after the operation and at week 4 and 12 after surgery
  This questionnaire is a well validated and commonly used self-report measure to assess the severity of pain and the interference of pain with daily activities as well as the quality of life, patient's subjective experience of disease and treatment. The BPI assesses pain at its "worst," "least," "average," and "now" (current pain) on a scale from 0 (no pain) to 10 (pain as bad as you can imagine) during the past 24 hours A clinically meaningful change in worst pain is defined as a change from baseline of at least 2 points in either direction. The BPI measures how much pain has interfered general activity, walking, work, mood, enjoyment of life, relations with others, and sleep. BPI pain interference is typically scored as the mean of the seven interference items. This mean can be used if more than 50% or four of seven of the total items have been completed on a given administration.
Patient Euro quality of life questionnaire (EQ-5D) | every day during the first 2 weeks after the operation and at week 4 and 12 after surgery
  EuroQol Group developed the questionnaire to describe and value health-related quality of life patient's subjective experience of disease and treatment. This includes 5 assessments: mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each assessment has 5 levels: no problems (1), slight problems (2), moderate problems (3), severe problems (4) and extreme problems (5). The patient ticks the box against the most appropriate statement in each of the 5 dimensions, which are summed in a 5-digit number describing the respondent's health state: having no problems for 1, slight problems for 2, moderate problems for 3, severe problems for 4 and extreme problems for 5.
  On the form there is also a scale with numbers from 0 to 100. 100 is the best health and 0 the worst health the patient can imagine. The patient has to tick the appropriate number.
Health Economic Analysis (HEA) | at week 4 and week 12
  forms are completed by the investigator and collect data on hospitalizations, rehabilitation, stays at nursing homes, out-patient visits performed by physicians working at practice offices or at hospitals, treatments as physiotherapy,nutrition counseling or alternative therapies

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Berclaz, Principal Investigator — Brustzentrum Bern
Locations (1):
- Brustzentrum Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The Clinical Trial Unit of the University of Bern will perform the statistical analysis and will be involved in the publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 3 years after study end
Access Criteria: 3 years after study end

REFERENCES:
- [Background] Kuroi K, Shimozuma K, Taguchi T, Imai H, Yamashiro H, Ohsumi S, Saito S. Effect of mechanical closure of dead space on seroma formation after breast surgery. Breast Cancer. 2006;13(3):260-5. doi: 10.2325/jbcs.13.260. PMID 16929119
- [Result] Barton A, Blitz M, Callahan D, Yakimets W, Adams D, Dabbs K. Early removal of postmastectomy drains is not beneficial: results from a halted randomized controlled trial. Am J Surg. 2006 May;191(5):652-6. doi: 10.1016/j.amjsurg.2006.01.037. PMID 16647354
- [Result] Tadych K, Donegan WL. Postmastectomy seromas and wound drainage. Surg Gynecol Obstet. 1987 Dec;165(6):483-7. PMID 3686312
- [Result] Tejler G, Aspegren K. Complications and hospital stay after surgery for breast cancer: a prospective study of 385 patients. Br J Surg. 1985 Jul;72(7):542-4. doi: 10.1002/bjs.1800720714. PMID 4016536
- [Result] Pogson CJ, Adwani A, Ebbs SR. Seroma following breast cancer surgery. Eur J Surg Oncol. 2003 Nov;29(9):711-7. doi: 10.1016/s0748-7983(03)00096-9. PMID 14602488
- [Result] Aitken DR, Minton JP. Complications associated with mastectomy. Surg Clin North Am. 1983 Dec;63(6):1331-52. doi: 10.1016/s0039-6109(16)43192-0. No abstract available. PMID 6359504
- [Result] Bryant M, Baum M. Postoperative seroma following mastectomy and axillary dissection. Br J Surg. 1987 Dec;74(12):1187. doi: 10.1002/bjs.1800741239. No abstract available. PMID 3427377
- [Result] Boostrom SY, Throckmorton AD, Boughey JC, Holifield AC, Zakaria S, Hoskin TL, Degnim AC. Incidence of clinically significant seroma after breast and axillary surgery. J Am Coll Surg. 2009 Jan;208(1):148-50. doi: 10.1016/j.jamcollsurg.2008.08.029. Epub 2008 Oct 2. No abstract available. PMID 19228516
- [Result] Kuroi K, Shimozuma K, Taguchi T, Imai H, Yamashiro H, Ohsumi S, Saito S. Pathophysiology of seroma in breast cancer. Breast Cancer. 2005;12(4):288-93. doi: 10.2325/jbcs.12.288. PMID 16286909
- [Result] Sampathraju S, Rodrigues G. Seroma formation after mastectomy: pathogenesis and prevention. Indian J Surg Oncol. 2010 Dec;1(4):328-33. doi: 10.1007/s13193-011-0067-5. Epub 2011 Apr 2. PMID 22693384
- [Result] Kumar S, Lal B, Misra MC. Post-mastectomy seroma: a new look into the aetiology of an old problem. J R Coll Surg Edinb. 1995 Oct;40(5):292-4. PMID 8523301
- [Result] Gonzalez EA, Saltzstein EC, Riedner CS, Nelson BK. Seroma formation following breast cancer surgery. Breast J. 2003 Sep-Oct;9(5):385-8. doi: 10.1046/j.1524-4741.2003.09504.x. PMID 12968958
- [Result] van Bemmel AJ, van de Velde CJ, Schmitz RF, Liefers GJ. Prevention of seroma formation after axillary dissection in breast cancer: a systematic review. Eur J Surg Oncol. 2011 Oct;37(10):829-35. doi: 10.1016/j.ejso.2011.04.012. Epub 2011 Aug 17. PMID 21849243
- [Result] Hashemi E, Kaviani A, Najafi M, Ebrahimi M, Hooshmand H, Montazeri A. Seroma formation after surgery for breast cancer. World J Surg Oncol. 2004 Dec 9;2:44. doi: 10.1186/1477-7819-2-44. PMID 15588301
- [Result] Aitken DR, Hunsaker R, James AG. Prevention of seromas following mastectomy and axillary dissection. Surg Gynecol Obstet. 1984 Apr;158(4):327-30. PMID 6369582
- [Result] Sakkary MA. The value of mastectomy flap fixation in reducing fluid drainage and seroma formation in breast cancer patients. World J Surg Oncol. 2012 Jan 11;10:8. doi: 10.1186/1477-7819-10-8. PMID 22236813
- [Result] Kopelman D, Klemm O, Bahous H, Klein R, Krausz M, Hashmonai M. Postoperative suction drainage of the axilla: for how long? Prospective randomised trial. Eur J Surg. 1999 Feb;165(2):117-20; discussion 121-2. doi: 10.1080/110241599750007289. PMID 10192568
- [Result] Porter KA, O'Connor S, Rimm E, Lopez M. Electrocautery as a factor in seroma formation following mastectomy. Am J Surg. 1998 Jul;176(1):8-11. doi: 10.1016/s0002-9610(98)00093-2. PMID 9683123
- [Result] Lumachi F, Brandes AA, Burelli P, Basso SM, Iacobone M, Ermani M. Seroma prevention following axillary dissection in patients with breast cancer by using ultrasound scissors: a prospective clinical study. Eur J Surg Oncol. 2004 Jun;30(5):526-30. doi: 10.1016/j.ejso.2004.03.003. PMID 15135481
- [Result] Burak WE Jr, Goodman PS, Young DC, Farrar WB. Seroma formation following axillary dissection for breast cancer: risk factors and lack of influence of bovine thrombin. J Surg Oncol. 1997 Jan;64(1):27-31. doi: 10.1002/(sici)1096-9098(199701)64:13.0.co;2-r. PMID 9040797
- [Result] Sanders RP, Goodman NC, Amiss LR Jr, Pierce RA, Moore MM, Marx G, Morgan RF, Spotnitz WD. Effect of fibrinogen and thrombin concentrations on mastectomy seroma prevention. J Surg Res. 1996 Feb 15;61(1):65-70. doi: 10.1006/jsre.1996.0082. PMID 8769944
- [Result] Medl M, Mayerhofer K, Peters-Engl C, Mahrhofer P, Huber S, Buxbaum P, Sevelda P, Leodolter S. The application of fibrin glue after axillary lymphadenectomy in the surgical treatment of human breast cancer. Anticancer Res. 1995 Nov-Dec;15(6B):2843-5. PMID 8669876
- [Result] Jain PK, Sowdi R, Anderson AD, MacFie J. Randomized clinical trial investigating the use of drains and fibrin sealant following surgery for breast cancer. Br J Surg. 2004 Jan;91(1):54-60. doi: 10.1002/bjs.4435. PMID 14716794
- [Result] Rice DC, Morris SM, Sarr MG, Farnell MB, van Heerden JA, Grant CS, Rowland CM, Ilstrup DM, Donohue JH. Intraoperative topical tetracycline sclerotherapy following mastectomy: a prospective, randomized trial. J Surg Oncol. 2000 Apr;73(4):224-7. doi: 10.1002/(sici)1096-9098(200004)73:43.0.co;2-0. PMID 10797336
- [Result] Chilson TR, Chan FD, Lonser RR, Wu TM, Aitken DR. Seroma prevention after modified radical mastectomy. Am Surg. 1992 Dec;58(12):750-4. PMID 1456600
- [Result] Ouldamer L, Caille A, Giraudeau B, Body G. Quilting Suture of Mastectomy Dead Space Compared with Conventional Closure with Drain. Ann Surg Oncol. 2015 Dec;22(13):4233-40. doi: 10.1245/s10434-015-4511-6. Epub 2015 Mar 18. PMID 25783681
- [Result] ten Wolde B, van den Wildenberg FJ, Keemers-Gels ME, Polat F, Strobbe LJ. Quilting prevents seroma formation following breast cancer surgery: closing the dead space by quilting prevents seroma following axillary lymph node dissection and mastectomy. Ann Surg Oncol. 2014 Mar;21(3):802-7. doi: 10.1245/s10434-013-3359-x. Epub 2013 Nov 12. PMID 24217790
- [Result] Coveney EC, O'Dwyer PJ, Geraghty JG, O'Higgins NJ. Effect of closing dead space on seroma formation after mastectomy--a prospective randomized clinical trial. Eur J Surg Oncol. 1993 Apr;19(2):143-6. PMID 8491318
- [Result] Ouldamer L, Trefoux-Bourdet A, Duquesne M, Body G. [How I do ... quilting suture of dead space after mastectomy]. Gynecol Obstet Fertil. 2011 Nov;39(11):663-4. doi: 10.1016/j.gyobfe.2011.07.041. Epub 2011 Oct 13. No abstract available. French. PMID 22000027
- [Result] Soon PS, Clark J, Magarey CJ. Seroma formation after axillary lymphadenectomy with and without the use of drains. Breast. 2005 Apr;14(2):103-7. doi: 10.1016/j.breast.2004.09.011. PMID 15767179
- [Result] Jeffrey SS, Goodson WH 3rd, Ikeda DM, Birdwell RL, Bogetz MS. Axillary lymphadenectomy for breast cancer without axillary drainage. Arch Surg. 1995 Aug;130(8):909-12; discussion 912-3. doi: 10.1001/archsurg.1995.01430080111018. PMID 7632155
- [Result] Gauthier T, Garuchet-Bigot A, Marin B, Mollard J, Loum O, Fermeaux V, Jammet I, Kanoun D, Maubon A, Aubard Y. Lanreotide Autogel 90 mg and lymphorrhea prevention after axillary node dissection in breast cancer: a phase III double blind, randomized, placebo-controlled trial. Eur J Surg Oncol. 2012 Oct;38(10):902-9. doi: 10.1016/j.ejso.2012.05.009. Epub 2012 Jun 15. PMID 22703757
- [Result] Shamley DR, Barker K, Simonite V, Beardshaw A. Delayed versus immediate exercises following surgery for breast cancer: a systematic review. Breast Cancer Res Treat. 2005 Apr;90(3):263-71. doi: 10.1007/s10549-004-4727-9. PMID 15830140
- [Result] Schuijtvlot M, Sahu AK, Cawthorn SJ. A prospective audit of the use of a buttress suture to reduce seroma formation following axillary node dissection without drains. Breast. 2002 Feb;11(1):94-6. doi: 10.1054/brst.2001.0366. PMID 14965653